CLINICAL TRIAL: NCT02204241
Title: A Multicenter, Open Label Phase I/II Study of Carfilzomib, Cyclophosphamide and Dexamethasone in Newly Diagnosed Multiple Myeloma (MM) Patients
Brief Title: Study of Carfilzomib, Cyclophosphamide and Dexamethasone in Newly Diagnosed Multiple Myeloma Patients
Acronym: CCD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Myeloma Network B.V. (Network)
Collaborators: Fondazione EMN Italy Onlus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IST-CAR-601
Record Dates: First submitted 2014-07-04; First posted 2014-07-30 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-05

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma; Diagnosis; CCyd
MeSH Terms: conditions — Multiple Myeloma; Disease | interventions — carfilzomib; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CCyd (Experimental): Treatment schedule for 9 cycles of induction:
  Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9,15-16, 22-23.
  Carfilzomib given 20 mg/m2 IV once daily on Day 1-2 of Cycle 1 only followed by 36/45/56/70 mg/m2 on days 8-9, 15-16 of Cycle 1, then for all subsequent doses 36/45/56/70 mg/m2 IV once daily on days 1-2, 8-9, 15-16, followed by 12-day rest period (day 17 through 28).
  Treatment schedule for maintenance until progression or intolerance:
  Carfilzomib at the MTD defined by phase I study IV once daily on days 1-2, 15-16.
  Interventions: Drug: Carfilzomib; Drug: Cyclophosphamide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Carfilzomib
Drug: Cyclophosphamide
Drug: Dexamethasone

SUMMARY:
This protocol is a phase I/II multicenter study designed to assess the safety and the efficacy of the proposed combinations as up-front treatment in elderly Multiple Myeloma (MM) patients.

DETAILED DESCRIPTION:
Treatment schedule for 9 cycles of induction:

Phase I:

In the phase I portion of the study, the following dose levels of carfilzomib will be studied with fixed doses of dexamethasone and cyclophosphamide to define the maximum tolerated dose (MTD):

Level-1:

1. Carfilzomib given 20 mg/m2 IV once daily on days 1-2 of Cycle 1 only followed by 36 mg/m2 on days 8-9, 15-16, of Cycle 1, then for all subsequent doses 36 mg/m2 IV once daily on days 1-2, 8-9, 15-16.
2. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15
3. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9, 15-16, 22-23

Level 0:

1. Carfilzomib given 20 mg/m2 IV once daily on days 1-2 of Cycle 1 only followed by 45 mg/m2 on days 8-9, 15-16, of Cycle 1, then for all subsequent doses 45 mg/m2 IV once daily on days 1-2, 8-9, 15-16.
2. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15
3. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9, 15-16, 22-23

Level +1:

1. Carfilzomib given 20 mg/m2 IV once daily on days 1-2 of Cycle 1 only followed by 56 mg/m2 on days 8-9, 15-16, of Cycle 1, then for all subsequent doses 56 mg/m2 IV once daily on days 1-2, 8-9, 15-16.
2. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15
3. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9, 15-16, 22-23

Level +2:

1. Carfilzomib given 20 mg/m2 IV once daily on days 1-2 of Cycle 1 only followed by 36 mg/m2 on days 8-9, 15-16, of Cycle 1, then for all subsequent doses 70 mg/m2 IV once daily on days 1-2, 8-9, 15-16.
2. Cyclophosphamide given orally at the dose of 300 mg/m2 on days 1, 8, 15
3. Dexamethasone given orally at the dose of 40 mg on days 1, 8, 15, 22 or 20 mg on days 1-2, 8-9, 15-16, 22-23

Patient will be observed at the end of the second cycle of therapy for the assessment of side effects and observation of DLTs. Dose escalation will proceed as follows:

* 3 patients will be entered at dose level 0
* If 0/3 patients experience DLT, dose escalation will continue
* If 1/3 patients experience DLT, 3 additional patients will be added to this cohort (max 6)
* If no further patients experience DLT (1/6) dose escalation will continue
* If 2/6 patients experience DLT, the MTD will have been exceeded and the MTD will be the previous dose at which <2/6 experienced DLT
* If 2/3 patients experience a DLT at any given dose, the MTD will have been exceeded and the MTD will be the preceding dose at which < 2/6 (or 1/3) patients experienced a DLT.

Phase II:

The dose used to treat patients in the phase II will be the MTD defined in the phase I of the study.

Treatment schedule for maintenance until progression or intolerance:

Carfilzomib at the MTD defined by phase I study IV once daily on days 1-2, 15-16.

ELIGIBILITY:
Inclusion Criteria:

* Patient is of a legally consenting age as defined by local regulations.
* Patient is age ≥ 65 year of age or who are ineligible for autologous stem cell transplantation.
* Patient is, in the investigator(s) opinion, willing and able to comply with the protocol requirements.
* Patient has given voluntary written informed consent before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to their future medical care.
* Women of childbearing potential must have a negative serum pregnancy test within the 7 days prior to study drug administration and a negative urine pregnancy test within the 3 days prior to the first study drug administration.
* Women of childbearing potential and male subjects who are sexullay active with WOCBP must agree to use 2 highly effective methods of contraception during the study and for 30 days following the last dose of study treatment including a male condom.
* Patient is a newly diagnosed MM patient.
* Patient has measurable disease, defined as follows: any quantifiable serum monoclonal protein value (generally, but not necessarily, ≥ 0.5 g/dL of M-protein) and, where applicable, urine light-chain excretion of >200 mg/24 hours. For patients with oligo or non-secretory MM, it is required that they have measurable plasmacytoma > 2 cm as determined by clinical examination or applicable radiographs (i.e. MRI, CT-Scan) or an abnormal free light chain ratio (n.v.: 0.26-1.65). We anticipate that less than 10% of patients admitted to this study will be oligo- or non-secretory MM with free light chains only in order to maximize interpretation of benefit results.
* Patient has a Karnofsky performance status ≥60%.
* Patient has a life-expectancy >3 months.
* Patient has the following laboratory values within 14 days before Baseline (day 1 of the Cycle 1, before study drug administration):

  * Platelet count ≥50 x 109/L (≥30 x 109 /L if myeloma involvement in the bone marrow is > 50%) within 14 days prior to drug administration.
  * Absolute neutrophil count (ANC) ≥ 1 x 109/L without the use of growth factors.
  * Corrected serum calcium ≤14 mg/dL (3.5 mmol/L)
  * Alanine transaminase (ALT): ≤ 3 x the ULN.
  * Total bilirubin: ≤ 2 x the ULN.
  * Calculated or measured creatinine clearance: ≥ 15 mL/minute
  * LVEF ≥40%. 2D transthoracic ECHO is the preferred method of evaluation. Multigated Acquisition Scan is acceptable if ECHO is not available

Exclusion Criteria:

* Patients with non-secretory MM, unless serum free light chains are present and the ratio is abnormal.
* Women who are pregnant and/or breast feeding.
* Patient has active infectious hepatitis type B or C or HIV.
* Pulmonary Hypertension.
* QTc Interval ≥ 450 msec.
* Uncontrolled Atrial Fibrillation/Flutter.
* History of Torsade de pointe, Ventricular Tachycardia, Ventricular Fibrillation.
* Uncontrolled Infection.
* Patients with myocardial infarction or unstable angina ≤ 4 months or other clinically significant heart disease (e.g., CHF NY Heart Association class III or IV, uncontrolled hypertension, history of labile hypertension, or history of poor compliance with an antihypertensive regimen).
* Patient with peripheral neuropathy > CTCAE grade 2.
* Known history of allergy to Captisol (a cyclodextrin derivative used to solubilize carfilzomib).
* Contraindication to any of the required concomitant drugs or supportive treatments, including hypersensitivity to all anticoagulation and antiplatelet options, antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment.
* Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to baseline.
* Patient has any other clinically significant illness that would, in the investigator's opinion, increase the patient's risk for toxicity.
* Patients with a prior malignancy within the last 5 years (except for basal or squamous cell carcinoma, or in situ cancer of the cervix or breast, or localized prostate cancer of Gleason score <7 with a stable PSA).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2023-04 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 1 year
  Non-hematologic:
  * Grade 2 neuropathy with pain
  * any Grade 3 tox. (excluding nausea, vomiting, diarrhea)
  * Grade 3 nausea, vomiting, or diarrhea despite maximal antiemetic/antidiarrheal therapy
  * Grade 4 fatigue lasting for ≥ 7 days
    * Any non-hematologic tox. requiring a dose reduction within Cycle 1
    * Inability to receive Day 1 dose of Cycle 2 due to drug related tox. persisting from Cycle 1 or drug related tox. newly encountered on Day 1 of Cycle 2.
  Hematologic:
  * Grade 4 neutropenia (ANC < 0.5 x 109/L) lasting for ≥ 7 days
  * Febrile neutropenia (ANC < 1.0 x 109/L with a fever ≥ 38.3ºC)
  * Grade 4 thrombocytopenia (platelets < 25.0 x 109/L) lasting ≥ 7 days despite dose delay
  * Grade 3-4 thrombocytopenia associated with bleeding
  * Any hematologic tox. requiring a dose reduction within Cycle 1
  * Inability to receive Day 1 dose of Cycle 2 due to drug related tox. persisting from Cycle 1 or drug related tox. newly encountered on Day 1 of Cycle 2.

SECONDARY OUTCOMES:
Response rate (RR) | 3 years
  Determine the response rate
Progression-free survival (PFS) | 3 years
  Determine the progression-free survival (PFS)
Time to progression (TTP) | 3 years
  Determine the time to progression (TTP)
Duration of response (DOR) | 3 years
  Determine the duration of response (DOR)
Overall survival (OS) | 3 years
  Determine the overall survival (OS)
Time to next therapy (TTNT) | 3 years
  Determine the time to next therapy (TTNT)
Responses | 3 years
  Determine whether responses obtained with CCyd treatment are associated with a prolongation of PFS, in comparison with non-responding patients
Response and survival | 3 years
  Determine whether tumor response and outcome may change in subgroups with different prognosis according to current prognostic factors (β2-microglobulin, C-reactive protein (CRP), FISH, gene expression profile)
Maintenance | 3 years
  Determine the benefit on PFS and OS of maintenance with carfilzomib
Adverse event | 1 years
  The toxicity is defined as the first occurrence of a grade 4 hematologic drug-related toxicity (grade 4 neutropenia must last longer than 3 days and grade 4 thrombocytopenia must last longer than 7 days in order to be considered a toxicity) excluding anemia. Assessment of adverse events will be performed at the end of third cycle according to the National Cancer Institute Common Terminology Criteria of Adverse Events (CTCAE version 4.0).

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione EMN Italy Onlus, Torino, Italy